CLINICAL TRIAL: NCT05193968
Title: Hot Flashes and Neurovascular Function in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sarah E. Baker, Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-002638; K01HL148144 (NIH)
Record Dates: First submitted 2021-11-15; First posted 2022-01-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Hot Flashes; Menopause; Vasomotor System; Labile
Keywords: Neurovascular function; Autonomic function; Microvascular Function
MeSH Terms: conditions — Hot Flashes | interventions — Valsalva Maneuver; Nitroprusside; Acetylcholine; Terbutaline; Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Healthy Women Volunteers (Other): Hot Flash frequency will be assessed in the study subjects during a screening period. Participants can then chose to participate 1 or 2 study visits- Protocol 1: Microvascular function and/or Protocol 2: Autonomic function
  Interventions: Other: Sympathoexcitatory stressors; Drug: Sodium Nitroprusside; Drug: Acetylcholine; Drug: Terbutaline; Drug: Norepinephrine

INTERVENTIONS:
Other: Sympathoexcitatory stressors — Muscle sympathetic nerve activity will be measured continuously at baseline and in response to sympathoexcitatory stressors, including a Valsalva maneuver, isometric handgrip exercise, a cold pressor test, and stepped hypercapnia.
  Other Names: Valsalva maneuver, handgrip exercise, ice water, and hypercapnia
Drug: Sodium Nitroprusside — Sodium nitroprusside, used to test endothelium-independent vasodilation, will be infused through a brachial artery catheter at 0.25, 0.5, 1.0 and 2.0 ug/100ml tissue/min.
  Other Names: Forearm vascular conductance response to sodium nitroprusside
Drug: Acetylcholine — Acetylcholine, used to test endothelium-dependent vasodilation, will be infused through a brachial artery catheter at 1.0, 2.0, 4.0, and 8.0 μg/100ml tissue/min
  Other Names: Forearm vascular conductance response to acetylcholine
Drug: Terbutaline — Terbutaline, a β2-Adrenergic selective agonist, will be infused through a brachial artery catheter at 0.1, 0.5, 1.0, and 2.0 μg/100ml tissue/min.
  Other Names: Forearm vascular conductance response to terbutaline
Drug: Norepinephrine — Norepinephrine, an α-adrenergic vasoconstricting agent, will be infused through a brachial artery catheter at 1.0, 2.0, 4.0, and 8.0 ng/100ml tissue/min
  Other Names: Forearm vascular conductance response to norepinephrine

SUMMARY:
Women who experience hot flashes are at greater risk for hypertension and other cardiovascular disease. Neurovascular control mechanisms are likely to play an important role in this relationship. As such, these studies are designed to provide a major step forward in understanding the link between hot flashes and neurovascular dysfunction and, by extension, cardiovascular disease in women.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers.
* Non-obese.
* Have at least one ovary.
* Free from cardiovascular disease.
* Not taking medications influencing cardiovascular function.

Exclusion Criteria:

- None.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-02-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Compare microvascular function in women with low and high frequency hot flashes | Continuous measurement of vascular conductance during infusion of each drug- 3min at baseline and at each drug dose (~60min total of continuous forearm vascular conductance measurements)
  Change in forearm vascular conductance with intra-arterial drug infusions.
  Vascular conductance is an index of vascular tone and is assessed using a technique called venous occlusion plethysmography
Compare sympathetic function in women with low and high frequency hot flashes | Continuous measurement of muscle sympathetic nerve activity at rest and in response to stressors (~75min of continuous data collection once a sympathetic nerve signal is found)
  Muscle Sympathetic Nerve Activity will be directly using a technique called microneurography.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Baker, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials